CLINICAL TRIAL: NCT04326647
Title: Short-term Effects Kinesiotaping (KT) on Balance and Gait in Parkinson's Disease (DP)
Acronym: KT-DP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jma002
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease; Kinesiotaping
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping Group (Experimental): We used kinesiotaping (gastrocnemius and lumbar back) plus exercise
  Interventions: Other: Kinesiotaping
- Exercise Group (Active Comparator): We used only exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Kinesiotaping — We used kinesiotaping in gastrocnemius and lumbar back
  Arms: Kinesiotaping Group
Other: Exercise — Exercises about balance and gait
  Arms: Exercise Group

SUMMARY:
To analyze the short-term effect of kinesiotaping in balance and gait on Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III PD, according to the Hoehn and Yahr scale.
* Subjects who are in the age range of 50 to 80 years.
* Acceptance of informed consent.
* Not present a musculoskeletal disorder or other neurological disease that interferes with balance and / or walking.
* Not having a diagnosed vestibular disorder.

Exclusion Criteria:

* Diagnosis of parkinsonism o Parkison-Like.
* Taking medications that may interfere with the different variables evaluated.
* Allergy to any component of the bandage.
* Being a pacemaker.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Berg Test - T0 | up to week
  Berg Test pre-intervention
Berg Test - T1 | up to week
  Berg Test post-intervention two days
Berg Test - T2 | up to week
  Berg Test post-intervention seven days
Tinetti Gait Test - T0 | up to week
  Tinetti Gait Test pre-intervention
Tinetti Gait Test - T1 | up to week
  Tinetti Gait Test post-intervention two days
Tinetti Gait Test - T2 | up to week
  Tinetti Gait Test post-intervention seven days
Up & Go Test - T0 | up to week
  Up & Go Test pre-intervention
Up & Go Test - T1 | up to week
  Up & Go Test post-intervention two days
Up & Go Test - T2 | up to week
  Up & Go Test post-intervention seven days
Parkinson's Disease Questionnaire - T0 | up to month
  Parkinson's Disease Questionnaire pre-intervention
Parkinson's Disease Questionnaire - T1 | up to month
  Parkinson's Disease Questionnaire post-intervention
surface electromyography -T0 | up to week
  surface electromyography pre-intervention
surface electromyography -T1 | up to week
  surface electromyography post-intervention two days
surface electromyography -T2 | up to week
  surface electromyography post-intervention seven days

CONTACTS AND LOCATIONS:
Locations (1):
- Javier Merino Andrés, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No